

# **Trial Statistical Analysis Plan**

c20741038-03

**BI Trial No.:** 1200.120 Title: Phase I/II open label, dose escalation trial to determine the MTD, safety, PK and efficacy of afatinib monotherapy in children aged ≥1 year to <18 years with recurrent/refractory neuroectodermal tumours, rhabdomyosarcoma and/or other solid tumours with known ErbB pathway deregulation regardless of tumour histology Including Protocol Amendment 1 (c02332639-03), 2 (c02332639-04) and 3 (c02332639-05) Giotrif®, Gilotrif®, Afatinib Capsules and Solvent for Oral **Investigational Product(s):** Solution Responsible trial statistician(s): Phone: Fax: **Date of statistical** 31 JUL 2020 REVISED analysis plan: Revised Version: **** 

Proprietary confidential information

© 2020 Boehringer Ingelheim International GmbH or one or more of its affiliated companies. All rights reserved.

This document may not - in full or in part - be passed on, reproduced, published or otherwise used without prior written permission.

TSAP for BI Trial No: 1200.120 

Proprietary confidential information © 2020 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 1. **TABLE OF CONTENTS**

| TITLE | PAGE | 1 |
|------------|------------------------------------------------|----|
| 1. | TABLE OF CONTENTS | 2 |
| LIST O | F TABLES | 4 |
| 2. | LIST OF ABBREVIATIONS | 5 |
| 3. | INTRODUCTION | 7 |
| 4. | CHANGES IN THE PLANNED ANALYSIS OF THE STUDY | 8 |
| 5. | ENDPOINT(S) | |
| 5.1 | PRIMARY ENDPOINT(S) | |
| 5.2 | SECONDARY ENDPOINT(S) | |
| 5.2.1 | Key secondary endpoint(s) | |
| 5.2.2 | Secondary endpoint(s) | |
| | CENTED AT ANALYSIS DEPONICACIONS | 10 |
| 6. | GENERAL ANALYSIS DEFINITIONS | |
| 6.1 | TREATMENT(S) | |
| 6.2 | IMPORTANT PROTOCOL DEVIATIONS | |
| 6.3 | PATIENT SETS ANALYSED | 15 |
| 6.5 | POOLING OF CENTRES | |
| 6.6 | HANDLING OF MISSING DATA AND OUTLIERS | 16 |
| <b>6.7</b> | BASELINE, TIME WINDOWS AND CALCULATED VISITS | 17 |
| 7. | PLANNED ANALYSIS | 18 |
| <b>7.1</b> | DEMOGRAPHIC AND OTHER BASELINE CHARACTERISTICS | 18 |
| 7.2 | CONCOMITANT DISEASES AND MEDICATION | 18 |
| 7.3 | TREATMENT COMPLIANCE | |
| 7.4 | PRIMARY ENDPOINT(S) | |
| 7.4.1 | Dose Finding Part: | |
| 7.4.2 | MTD expansion cohort part: | |
| 7.5 | SECONDARY ENDPOINT(S) | |
| 7.5.1 | Key secondary endpoint(s) | |
| 7.5.2 | (Other) Secondary endpoint(s) | |
| 7.7 | EXTENT OF EXPOSURE | 20 |
| 7.8 | SAFETY ANALYSIS | |
| 7.8.1 | Adverse events | |
| 7.8.2 | Laboratory data | |
| 7.8.3 | Vital signs. | |
| 7.8.4 | ECG. | |
| 7.8.5 | Others | |
| 8. | REFERENCES | |
| U. | NEFERENCES | 43 |

| Boehringer | Ingelheim |
|------------|-----------|

| TSAP fo | r BI Trial No: 1200.120 | <b></b> |
|---|---|---|
| Proprietary c | onfidential information © 2020 Boehringer Ingelheim International GmbH or one or | more of its affiliated companies |
| 10. | HISTORY TABLE | 27 |

# **Boehringer Ingelheim**

TSAP for BI Trial No: 1200.120 
Proprietary confidential information © 2020 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

# LIST OF TABLES

| Table 6.1: 1 Definition of analysing treatment periods | |
|------------------------------------------------------------|----|
| Table 6.2: 1 Important protocol deviations | 1- |
| Table 7.4.2: 1 Confirmation rule for best overall response | |
| Table 7.8.2: 1 Primary laboratory parameters | 23 |
| Table 7.8.2: 2 Secondary laboratory parameters | 24 |
| Table 10: 1 History table | 27 |

TSAP for BI Trial No: 1200.120 
Proprietary confidential information © 2020 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 2. LIST OF ABBREVIATIONS

| AE Adverse event AUC Area Under Curve BMI Body mass index BRPM Blinded report planning meeting BSA Body surface area BUN Blood urea nitrogen Cmax Maximum Concentration CR Complete Response CTC Common Terminology Criteria CTP Clinical Trial Protocol CTR Clinical Trial Report DLT Dose Limiting Toxicity DM&SM Boehringer Ingelheim Data Management and Statistics Manual DoR Duration of objective response DRA Drug Regulatory Affairs EMA European Medicines Agency FAS Full analysis set FDA Food and Drug Administration ICH International Conference on Harmonisation INRC International Criteria for Neuroblastoma Response Criteria IPD Important protocol deviation LVEF Left ventricular ejection function MedDRA Medical Dictionary for Regulatory Activities MQRM Medical Quality Review Meeting MTD Maximum Tolerated Dose MxR Mixed response NOR Not-valid results NOS No sample available NR No response O*C Oracle Chincal | Term | Definition / description |
|---|---|---|
| BMI Body mass index BRPM Blinded report planning meeting BSA Body surface area BUN Blood urea nitrogen Cmax Maximum Concentration CR Complete Response CTC Common Terminology Criteria CTP Clinical Trial Protocol CTR Clinical Trial Report DLT Dose Limiting Toxicity DM&SM Boehringer Ingelheim Data Management and Statistics Manual DOR Duration of objective response DRA Drug Regulatory Affairs EMA European Medicines Agency FAS Full analysis set FDA Food and Drug Administration ICH International Conference on Harmonisation INRC International Criteria for Neuroblastoma Response Criteria IPD Important protocol deviation LVEF Left ventricular ejection function MedDRA Medical Dictionary for Regulatory Activities MQRM Medical Quality Review Meeting MTD Maximum Tolerated Dose MxR Mixed response NOR Not-valid results NOS No sample available NR No response O*C Oracle Clinical | AE | Adverse event |
| BRPM Blinded report planning meeting BSA Body surface area BUN Blood urea nitrogen Cmax Maximum Concentration CR Complete Response CTC Common Terminology Criteria CTP Clinical Trial Protocol CTR Clinical Trial Report DLT Dose Limiting Toxicity DM&SM Bochringer Ingelheim Data Management and Statistics Manual DOR Duration of objective response DRA Drug Regulatory Affairs EMA European Medicines Agency FAS Full analysis set FDA Food and Drug Administration ICH International Conference on Harmonisation INRC International Criteria for Neuroblastoma Response Criteria IPD Important protocol deviation LVEF Left ventricular ejection function MedDRA Medical Dictionary for Regulatory Activities MQRM Medical Quality Review Meeting MTD Maximum Tolerated Dose MxR Mixed response NOR Not-valid results NOS No sample available NR No response O*C Oracle Clinical | AUC | Area Under Curve |
| BSA Body surface area BUN Blood urea nitrogen Cmax Maximum Concentration CR Complete Response CTC Common Terminology Criteria CTP Clinical Trial Protocol CTR Clinical Trial Report DLT Dose Limiting Toxicity DM&SM Bochringer Ingelheim Data Management and Statistics Manual DOR Duration of objective response DRA Drug Regulatory Affairs EMA European Medicines Agency FAS Full analysis set FDA Food and Drug Administration ICH International Conference on Harmonisation INRC International Criteria for Neuroblastoma Response Criteria IPD Important protocol deviation LVEF Left ventricular ejection function MedDRA Medical Dictionary for Regulatory Activities MQRM Medical Quality Review Meeting MTD Maximum Tolerated Dose MxR Mixed response NOR Not-valid results NOS No sample available NR No response O*C Oracle Clinical | BMI | Body mass index |
| BUN Blood urea nitrogen Cmax Maximum Concentration CR Complete Response CTC Common Terminology Criteria CTP Clinical Trial Protocol CTR Clinical Trial Report DLT Dose Limiting Toxicity DM&SM Bochringer Ingelheim Data Management and Statistics Manual DOR Duration of objective response DRA Drug Regulatory Affairs EMA European Medicines Agency FAS Full analysis set FDA Food and Drug Administration ICH International Conference on Harmonisation INRC International Criteria for Neuroblastoma Response Criteria IPD Important protocol deviation LVEF Left ventricular ejection function MedDRA Medical Dictionary for Regulatory Activities MQRM Medical Quality Review Meeting MTD Maximum Tolerated Dose MxR Mixed response NOR Not-valid results NOS No sample available NR No response O*C Oracle Clinical | BRPM | Blinded report planning meeting |
| Cmax Maximum Concentration CR Complete Response CTC Common Terminology Criteria CTP Clinical Trial Protocol CTR Clinical Trial Report DLT Dose Limiting Toxicity DM&SM Boehringer Ingelheim Data Management and Statistics Manual DoR Duration of objective response DRA Drug Regulatory Affairs EMA European Medicines Agency FAS Full analysis set FDA Food and Drug Administration ICH International Conference on Harmonisation INRC International Criteria for Neuroblastoma Response Criteria IPD Important protocol deviation LVEF Left ventricular ejection function MedDRA Medical Dictionary for Regulatory Activities MQRM Medical Quality Review Meeting MTD Maximum Tolerated Dose MxR Mixed response NOR Not-valid results NOS No sample available NR No response O*C Oracle Clinical | BSA | Body surface area |
| CR Complete Response CTC Common Terminology Criteria CTP Clinical Trial Protocol CTR Clinical Trial Report DLT Dose Limiting Toxicity DM&SM Boehringer Ingelheim Data Management and Statistics Manual DoR Duration of objective response DRA Drug Regulatory Affairs EMA European Medicines Agency FAS Full analysis set FDA Food and Drug Administration ICH International Conference on Harmonisation INRC International Criteria for Neuroblastoma Response Criteria IPD Important protocol deviation LVEF Left ventricular ejection function MedDRA Medical Dictionary for Regulatory Activities MQRM Medical Quality Review Meeting MTD Maximum Tolerated Dose MxR Mixed response NOR Not-valid results NOS No sample available NR No response O*C Oracle Clinical | BUN | Blood urea nitrogen |
| CTC Common Terminology Criteria CTP Clinical Trial Protocol CTR Clinical Trial Report DLT Dose Limiting Toxicity DM&SM Boehringer Ingelheim Data Management and Statistics Manual DoR Duration of objective response DRA Drug Regulatory Affairs EMA European Medicines Agency FAS Full analysis set FDA Food and Drug Administration ICH International Conference on Harmonisation INRC International Criteria for Neuroblastoma Response Criteria IPD Important protocol deviation LVEF Left ventricular ejection function MedDRA Medical Dictionary for Regulatory Activities MQRM Medical Quality Review Meeting MTD Maximum Tolerated Dose MxR Mixed response NOR Not-valid results NOS No sample available NR No response O*C Oracle Clinical | $C_{max}$ | Maximum Concentration |
| CTP Clinical Trial Protocol CTR Clinical Trial Report DLT Dose Limiting Toxicity DM&SM Boehringer Ingelheim Data Management and Statistics Manual DoR Duration of objective response DRA Drug Regulatory Affairs EMA European Medicines Agency FAS Full analysis set FDA Food and Drug Administration ICH International Conference on Harmonisation INRC International Criteria for Neuroblastoma Response Criteria IPD Important protocol deviation LVEF Left ventricular ejection function MedDRA Medical Dictionary for Regulatory Activities MQRM Medical Quality Review Meeting MTD Maximum Tolerated Dose MxR Mixed response NOR Not-valid results NOS No sample available NR No response O*C Oracle Clinical | CR | Complete Response |
| CTR Clinical Trial Report DLT Dose Limiting Toxicity DM&SM Boehringer Ingelheim Data Management and Statistics Manual DoR Duration of objective response DRA Drug Regulatory Affairs EMA European Medicines Agency FAS Full analysis set FDA Food and Drug Administration ICH International Conference on Harmonisation INRC International Criteria for Neuroblastoma Response Criteria IPD Important protocol deviation LVEF Left ventricular ejection function MedDRA Medical Dictionary for Regulatory Activities MQRM Medical Quality Review Meeting MTD Maximum Tolerated Dose MxR Mixed response NOR Not-valid results NOS No sample available NR No response O*C Oracle Clinical | CTC | Common Terminology Criteria |
| DLT Dose Limiting Toxicity DM&SM Boehringer Ingelheim Data Management and Statistics Manual DoR Duration of objective response DRA Drug Regulatory Affairs EMA European Medicines Agency FAS Full analysis set FDA Food and Drug Administration ICH International Conference on Harmonisation INRC International Criteria for Neuroblastoma Response Criteria IPD Important protocol deviation LVEF Left ventricular ejection function MedDRA Medical Dictionary for Regulatory Activities MQRM Medical Quality Review Meeting MTD Maximum Tolerated Dose MxR Mixed response NOR Not-valid results NOS No sample available NR No response O*C Oracle Clinical | CTP | Clinical Trial Protocol |
| DM&SM Boehringer Ingelheim Data Management and Statistics Manual DOR Duration of objective response DRA Drug Regulatory Affairs EMA European Medicines Agency FAS Full analysis set FDA Food and Drug Administration ICH International Conference on Harmonisation INRC International Criteria for Neuroblastoma Response Criteria IPD Important protocol deviation LVEF Left ventricular ejection function MedDRA Medical Dictionary for Regulatory Activities MQRM Medical Quality Review Meeting MTD Maximum Tolerated Dose MxR Mixed response NOR Not-valid results NOS No sample available NR No response O*C Oracle Clinical | CTR | Clinical Trial Report |
| DoR Duration of objective response DRA Drug Regulatory Affairs EMA European Medicines Agency FAS Full analysis set FDA Food and Drug Administration ICH International Conference on Harmonisation INRC International Criteria for Neuroblastoma Response Criteria IPD Important protocol deviation LVEF Left ventricular ejection function MedDRA Medical Dictionary for Regulatory Activities MQRM Medical Quality Review Meeting MTD Maximum Tolerated Dose MxR Mixed response NOR Not-valid results NOS No sample available NR No response O*C Oracle Clinical | DLT | Dose Limiting Toxicity |
| DRA Drug Regulatory Affairs EMA European Medicines Agency FAS Full analysis set FDA Food and Drug Administration ICH International Conference on Harmonisation INRC International Criteria for Neuroblastoma Response Criteria IPD Important protocol deviation LVEF Left ventricular ejection function MedDRA Medical Dictionary for Regulatory Activities MQRM Medical Quality Review Meeting MTD Maximum Tolerated Dose MxR Mixed response NOR Not-valid results NOS No sample available NR No response O*C Oracle Clinical | DM&SM | Boehringer Ingelheim Data Management and Statistics Manual |
| EMA European Medicines Agency FAS Full analysis set FDA Food and Drug Administration ICH International Conference on Harmonisation INRC International Criteria for Neuroblastoma Response Criteria IPD Important protocol deviation LVEF Left ventricular ejection function MedDRA Medical Dictionary for Regulatory Activities MQRM Medical Quality Review Meeting MTD Maximum Tolerated Dose MxR Mixed response NOR Not-valid results NOS No sample available NR No response O*C Oracle Clinical | DoR | Duration of objective response |
| FAS Full analysis set FDA Food and Drug Administration ICH International Conference on Harmonisation INRC International Criteria for Neuroblastoma Response Criteria IPD Important protocol deviation LVEF Left ventricular ejection function MedDRA Medical Dictionary for Regulatory Activities MQRM Medical Quality Review Meeting MTD Maximum Tolerated Dose MxR Mixed response NOR Not-valid results NOS No sample available NR No response O*C Oracle Clinical | DRA | Drug Regulatory Affairs |
| FDA Food and Drug Administration ICH International Conference on Harmonisation INRC International Criteria for Neuroblastoma Response Criteria IPD Important protocol deviation LVEF Left ventricular ejection function MedDRA Medical Dictionary for Regulatory Activities MQRM Medical Quality Review Meeting MTD Maximum Tolerated Dose MxR Mixed response NOR Not-valid results NOS No sample available NR No response O*C Oracle Clinical | EMA | European Medicines Agency |
| ICH International Conference on Harmonisation INRC International Criteria for Neuroblastoma Response Criteria IPD Important protocol deviation LVEF Left ventricular ejection function MedDRA Medical Dictionary for Regulatory Activities MQRM Medical Quality Review Meeting MTD Maximum Tolerated Dose MxR Mixed response NOR Not-valid results NOS No sample available NR No response O*C Oracle Clinical | FAS | Full analysis set |
| INRC International Criteria for Neuroblastoma Response Criteria IPD Important protocol deviation LVEF Left ventricular ejection function MedDRA Medical Dictionary for Regulatory Activities MQRM Medical Quality Review Meeting MTD Maximum Tolerated Dose MxR Mixed response NOR Not-valid results NOS No sample available NR No response O*C Oracle Clinical | FDA | Food and Drug Administration |
| IPD Important protocol deviation LVEF Left ventricular ejection function MedDRA Medical Dictionary for Regulatory Activities MQRM Medical Quality Review Meeting MTD Maximum Tolerated Dose MxR Mixed response NOR Not-valid results NOS No sample available NR No response O*C Oracle Clinical | ICH | International Conference on Harmonisation |
| LVEF Left ventricular ejection function MedDRA Medical Dictionary for Regulatory Activities MQRM Medical Quality Review Meeting MTD Maximum Tolerated Dose MxR Mixed response NOR Not-valid results NOS No sample available NR No response O*C Oracle Clinical | INRC | International Criteria for Neuroblastoma Response Criteria |
| MedDRA Medical Dictionary for Regulatory Activities MQRM Medical Quality Review Meeting MTD Maximum Tolerated Dose MxR Mixed response NOR Not-valid results NOS No sample available NR No response O*C Oracle Clinical | IPD | Important protocol deviation |
| MQRM Medical Quality Review Meeting MTD Maximum Tolerated Dose MxR Mixed response NOR Not-valid results NOS No sample available NR No response O*C Oracle Clinical | LVEF | Left ventricular ejection function |
| MTD Maximum Tolerated Dose MxR Mixed response NOR Not-valid results NOS No sample available NR No response O*C Oracle Clinical | MedDRA | Medical Dictionary for Regulatory Activities |
| MxRMixed responseNORNot-valid resultsNOSNo sample availableNRNo responseO*COracle Clinical | MQRM | Medical Quality Review Meeting |
| NOR Not-valid results NOS No sample available NR No response O*C Oracle Clinical | MTD | Maximum Tolerated Dose |
| NOS No sample available NR No response O*C Oracle Clinical | MxR | Mixed response |
| NR No response O*C Oracle Clinical | NOR | Not-valid results |
| O*C Oracle Clinical | NOS | No sample available |
| | NR | No response |
| | O*C | Oracle Clinical |
| OR Objective Response | OR | Objective Response |

TSAP for BI Trial No: 1200.120 Proprietary confidential information © 2020 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

| Term | Definition / description |
|-----------|-------------------------------------|
| PD | Progressive Disease |
| PFS | Progression free survival |
| PK | Pharmacokinetics |
| PopPK | Population Pharmacokinetic(s) |
| PPS | Per protocol set |
| PPSR | Proposed pediatric study request |
| PR | Partial Response |
| PSTAT | Project Statistician |
| PT | Preferred term |
| Q1 | Lower quartile |
| Q3 | Upper quartile |
| SAS | Statistical Analysis System |
| s.d. | Standard deviation |
| SD | Stable Disease |
| SMQ | Standardised MedDRA query |
| SOC | System Organ Class |
| $t_{max}$ | Time to reach maximum concentration |
| TCM | Trial Clinical Monitor |
| TMW | Trial Medical Writer |
| TOC | Table of contents |
| TSAP | Trial Statistical Analysis Plan |
| TSTAT | Trial Statistician |
| VGPR | Very good partial response |

TSAP for BI Trial No: 1200.120

Proprietary confidential information © 2020 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

# 3. INTRODUCTION

As per ICH E9 (1), the purpose of this document is to provide a more technical and detailed elaboration of the principal features of the analysis described in the protocol and its amendments, and to include detailed procedures for executing the statistical analysis of the primary and secondary variables and other data.

This Trial Statistical Analysis Plan (TSAP) assumes familiarity with the Clinical Trial Protocol (CTP), including Protocol Amendments. In particular, the TSAP is based on the planned analysis specification as written in CTP Section 7 "Statistical Methods and Determination of Sample Size". Therefore, TSAP readers may consult the CTP for more background information on the study, e.g., on study objectives, study design and population, treatments, definition of measurements and variables, planning of sample size, randomization.

SAS® Version 9.4 will be used for all analyses.

TSAP for BI Trial No: 1200.120

Proprietary confidential information © 2020 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

# 4. CHANGES IN THE PLANNED ANALYSIS OF THE STUDY

The clinical trial protocol (CTP) v3 was amended based on the feedback received from the FDA during a PPSR request. The MTD expansion cohorts will now recruit up to 38 patients evaluable for OR based on biomarker selection criteria as well as specific tumour indications.

The definition of duration of objective response was misspecified in the CTP as the interval between the date of randomization and the earliest date of disease progression. The correct definition is clarified in Section 5.2.2 of this TSAP as the time from first documented response of CR, VGPR, PR, or MxR until the earliest of disease progression or death among patients with objective response.

#### **5. ENDPOINT(S)**

#### 5.1 PRIMARY ENDPOINT(S)

## Dose finding part:

- The primary endpoint is the **dose limiting toxicity** (DLT) measured during the first course of treatment. DLTs are defined in Table 4.1.4.1.2 of the CTP.
- Pharmacokinetics (AUC<sub> $\tau$ ,ss</sub>, C<sub>max,ss</sub>)

The primary objective of the dose finding part is to determine the maximum tolerated dose (MTD) of the study drug as defined by patients with DLT in a paediatric population. The MTD will be determined as the highest dose at which no more than 1/6 patients experienced DLT. The MTD evaluation period is defined as the initial 28 days of study treatment. Patients who developed DLT at any time during the initial 28 treatment days and patients who have completed the MTD evaluation period without missing more than 25% of the afatinib doses regardless of the reason will be referred to as patients evaluable for DLT.

# MTD expansion cohort part:

Objective response (OR) by investigator assessment according to the institutional response evaluation criteria for the given tumour type, assessed every 8 weeks until progression of disease.

#### 5.2 **SECONDARY ENDPOINT(S)**

#### 5.2.1 **Key secondary endpoint(s)**

There were no key secondary endpoints for this study.

#### 5.2.2 **Secondary endpoint(s)**

### Dose finding part:

- Objective response (OR) assessed by investigator according to the institutional response evaluation criteria for the given tumour type, assessed every 8 weeks until progression of disease
- **Pharmacokinetics** (AUC<sub>0-24</sub>, C<sub>max</sub>, t<sub>max(.ss)</sub> and accumulation (or effective) half-life)

### MTD expansion cohort part:

- **Progression free survival** (PFS) is defined as the duration of time from the date of first drug administration to the date of the first documented disease progression evaluated according to institutional response criteria or to the date of death from any cause, whichever occurs first. Censoring rules and dates of outcome for PFS under difference scenarios are specified in Table 5.2.2: 1.
- **Duration of objective response** (DoR) is defined as the time from first documented response of CR, VGPR, PR, or MxR until the earliest of disease progression or death among patients with objective response. Censoring rules and dates of outcomes follow the same specifications as for PFS in Table 5.2.2: 1 for applicable scenarios.
- **Pharmacokinetics** (AUC<sub> $\tau$ (,ss)</sub>, C<sub>max(,ss)</sub>, t<sub>max(,ss)</sub> and accumulation (or effective) half-life)

TSAP for BI Trial No: 1200.120 Proprietary confidential information © 2020 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

Censoring rules and determination of date of event or censoring for Table 5.2.2: 1 **PFS** 

| Situation | Outcome<br>(event or | Date of outcome |
|---|---|---|
| | censored) | |
| No baseline radiological assessment (no | censored | Date of first treatment administration |
| death before second scheduled | | |
| radiological assessment) | | |
| Death without progression. At most one | event | Date of death |
| missed radiological assessments, i.e. at | | |
| most 112 days between death and last | | |
| assessment (or treatment start date if no | | |
| post-baseline assessments). | | |
| Death without progression. Two or | censored | Date of last radiological assessment / |
| more missed radiological assessments, | | Date of first treatment administration |
| i.e. longer than 112 days between death | | if no post-baseline assessments |
| and last assessment (or treatment start | | |
| date if no post-baseline assessments). | | |
| No radiological assessment performed | censored | Date of first treatment administration |
| post-baseline, vital status is unknown or | | |
| patient is known to be alive | | |
| Progressed according to radiological | event | Date of radiological assessment of |
| assessment. At most one missed | | progression |
| radiological assessments, i.e. at most | | |
| 112 days between progression and last | | |
| assessment before progression. | | |
| Progressed according to radiological | censored | Date of last radiological assessment |
| assessment, i.e. longer than 112 days | | before progression |
| between progression and last | | |
| assessment before progression. | | |
| Alive and not progressed (irrespective | censored | Date of last radiological assessment |
| of missed radiological assessments) | | |
| Initiation of subsequent anti-cancer therapy | | |
| Subsequent anti-cancer therapy started | censored | Date of last radiological assessment |
| before progression or death | | before subsequent anti-cancer therapy |
| No baseline and/or post-baseline | censored | Date of first treatment administration |
| imaging and subsequent anti-cancer | | |
| therapy started prior to a death | | |
| 1 | | |

For further details on endpoints, please see CTP Section 5.

# **Boehringer Ingelheim**

TSAP for BI Trial No: 1200.120 Proprietary confidential information © 2020 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

# **Boehringer Ingelheim**

TSAP for BI Trial No: 1200.120 Proprietary confidential information © 2020 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

# 6. GENERAL ANALYSIS DEFINITIONS

# 6.1 TREATMENT(S)

Daily single oral doses of afatinib will be investigated in this study for paediatric patients. Dose escalation starts at 80% of the adult MTD by m<sup>2</sup> BSA and allometric scaling (Level 0) and can be escalated to 100% (level 1), 125% (level 2) and 150% (level 3) of the adult dose if required. In case level 0 exceeds the MTD, a dose level -1 will allow de-escalation to 50% of the adult MTD dose by m<sup>2</sup> BSA and allometric scaling. Oral solution is available for younger children and patients who cannot swallow afatinib film coated tablets.

Analysing treatment periods are defined in Table 6.1: 1 for reporting of treatment emergent AEs and safety laboratory data. An adverse event will be assigned to the analysing period where start date  $\leq$  onset date of AE < stop date.

Table 6.1: 1 Definition of analysing treatment periods

| Analysing treatment period | Start date (including) | Stop date (excluding) |
|---|---|---|
| Screening | Date of informed consent | Date of first intake of study drug |
| Course 1 | Date of first intake of study drug | Start date of Course 2, or date of first intake of study drug + 28 days if the patient did not start Course 2 |
| On-treatment | Date of first intake of study drug | Date of last intake of study drug + 29 days |
| Residual effect<br>period (REP) | Date of last intake of study drug<br>+ 1 day | Date of last intake of study drug + 29 day |
| Off-treatment | Date of last intake of study drug<br>+ 29 day | Date of last follow up visit + 1 day or date of death + 1 day whichever occurred first |

The residual effect period (REP) for afatinib is 28 days after last intake of afatinib. Data recorded between the first study drug intake until up to 28 days after the last study drug intake will be considered as on-treatment.

#### 6.2 IMPORTANT PROTOCOL DEVIATIONS

A protocol deviation is important if it affects the rights or safety of the study patients, or if it can potentially influence the primary outcome measurements in a non-negligible way. Patients with important protocol deviations (IPDs) that could potentially impact the evaluation of the primary endpoint(s) will be excluded.

The different categories of IPDs are defined in Table 6.2: 1. IPDs will be reviewed at Medical Quality Review Meetings (MQRMs) conducted periodically during the trial. A list of protocol deviations will be discussed at the report planning meetings (RPMs). If the data show other IPDs, this table will be supplemented accordingly at MQRMs or RPMs or through team review of the protocol deviation log. The decision whether a patient will be excluded from the analysis will be made at the final RPM prior to DBL.

Table 6.2: 1 Important protocol deviations

| Category/<br>Code | | Description | Comment/Example | Excluded from | Manual/<br>Automatic |
|---|---|---|---|---|---|
| A | | Inclusion/Exclusion Criteria | | | |
| | A1 | | | | |
| | A1.1 | Laboratories measurements | Exclusion criteria13,14,15 | None | Automatic |
| | A1.2 | Forbidden concomitant diagnoses | Exclusion criteria 4,5,7,9,10,11,12 | None | Automatic |
| | A1.3 | Female patients who are pregnant or doing breast feeding at baseline | Exclusion criteria 6 | None | Automatic |
| | A1.4 | Prohibited concomitant medications, radiotherapy and surgery | Exclusion criteria 1,2,3, 8 | None | Automatic |
| | A2 | | | | Automatic |
| | A2.1 | Patient does not have trial diagnosis | Inclusion criteria 1 | None | Automatic |
| | A2.2 | Patient did not recover (to CTCAE grade 1 or baseline) from any acute toxicity resulting from prior anti-cancer treatment (except alopecia) | Inclusion criteria 4 | None | Automatic |
| | A2.3 | Patient did not have Lansky/Karnofsky (depending on age) scores >=50% assessed within 2 weeks prior to enrolment. | Inclusion criteria 8 | None | Automatic |
| | A2.4 | Patient has LVEF <50% | Inclusion criteria 12 | None | Automatic |
| | A2.5 | Required ErbB pathway deregulation absent | MTD Expansion<br>Cohort: Inclusion<br>criteria 1 or 13 | None | Automatic |
| | A2.6 | Patient age at study start not between >=2 to <18 years | Dose finding cohort:<br>Inclusion criteria 3 | None | Automatic |
| | | Patient age at study start not between >=1 to <18 years | MTD expansion cohort: Inclusion criteria 3 | | |
| | A2. 7 | No tumour tissue available (exception of DIPG) | MTD Expansion<br>Cohort: Inclusion<br>criteria 7 | None | Automatic |
| | A2.8 | Patient do not have at least one measurable lesion according to the institutional response criteria for the given tumour type. | Inclusion criteria 14 | None | Automatic |

Table 6.2: 1 Important protocol deviations (cont.)

| | tegory/<br>Code | Description | Comment/Example | Excluded from | Manual/<br>Automatic |
|---|---|---|---|---|---|
| В | | Informed Consent | | | Automatic |
| | B1 | Informed consent not given | Inclusion criterion 6 | All | Automatic |
| | B2 | Informed consent after administration of trial medication | Inclusion criterion 6 | None | Automatic |
| | В3 | Informed consent not in accordance with regulations | | None | Manual |
| C | | Trial Medication | | | |
| | C1 | Dose change of afatinib not according to protocol | | None | Manual |
| | C2 | Non-compliance | Afatinib not taken according to protocol | None | Manual |
| | C3 | Dose reduction/paused/discontinuation not according to protocol following an AE/DLT | Refer to Table<br>4.1.2.3:1 and Table<br>4.2.2.1:1 in the CTP | None | Manual |
| D | | Concomitant Treatment | | | |
| | D1 | Any other chemotherapy, immunotherapy or radiotherapy during the trial except for palliative radiation | Refer to Section 4.2 of the CTP | None | Manual |
| | D2 | During palliative radiation, treatment was<br>not paused until the patient recovered from<br>any radiation associated toxicity | Refer to Section 4.2 of the CTP | None | Manual |
| | D3 | Continuous interruption of >28 days due to palliative radiotherapy | Refer to Section 4.2 of the CTP | None | Manual |
| Е | | Critical study procedure | | | |
| | E1 | Critical study procedure not followed | | None | Manual |
| F | | Privacy / data protection | | | |
| | F1 | Privacy and/or data protection violated | | None | Manual |

# 6.3 PATIENT SETS ANALYSED

# Treated set (TS):

This patient set includes all patients enrolled in the trial who were documented to have taken at least one dose of study medication.

# Dose finding cohort treated set:

This patient set includes all patients enrolled in dose finding cohort of the trial who were documented to have taken at least one dose of study medication.

## MTD Expansion cohort treated set:

This patient set includes all patients enrolled in expansion cohort who must satisfy the following criterion:

 Patients' tumour must be tested for positivity on 2 of the following tests: EGFR IHC>150 and/or HER2 IHC>0 and/or EGFR FISH positive and/or HER2 DDISH positive.

or

 Patient will have proven genomic, transcriptomic or proteomic alterations which are not defined above.

and

• Patients who were documented to have taken at least one dose of study medication.

#### PK analysis set (PKS):

This set includes all patients in the treated set (TS) who provided at least one PK endpoint that was not excluded due to a protocol deviation relevant to the evaluation of PK or due to PK non-evaluability. Thus, a patient will be included in the PKS, even if he/she contributes only one PK parameter value for one period to the statistical assessment. Descriptive and model based analyses of PK parameters will be based on the PKS.

#### 6.5 POOLING OF CENTRES

This section is not applicable.

#### 6.6 HANDLING OF MISSING DATA AND OUTLIERS

Missing or incomplete AE dates are imputed according to BI standards (3). Missing efficacy data, including vital status, tumour imaging data, will not be imputed in general. All reasonable efforts have been undertaken during the study to obtain such data.

Missing or incomplete drug stop dates are imputed as follows:

- If month and year known for drug stop date but day missing, then use date of death if within the month; otherwise use last day of month.
- If both month and day unknown, then use the first available date in this order: date of death, date of last contact, last day of the month of last visit.

Missing data and outliers of PK data are handled according to (2). Samples marked as no sample available (NOS) or non-valid result (NOR) will not be included in the analysis. Please refer to Sections 7.3.5 and 7.4 of the CTP for more details.

### 6.7 BASELINE, TIME WINDOWS AND CALCULATED VISITS

Study days and visits will be labelled according to the flow chart of the CTP. Unless otherwise specified, baseline is defined as the latest time point before the very first administration of any study medication. If this criterion is not fulfilled, then no baseline will be derived. Note that for some trial procedures (for example performance score, body weight, vital signs, laboratory tests) this may be the value measured on the same day when trial medication was started. In these cases it will be assumed that the measurements were taken prior to the intake of any study medication. For laboratory values where not only the examination date but also time are recorded, examination time has to be taken into account when defining baseline. That is, a laboratory value on the same date as the first study drug administration is considered as baseline value if and only if the time of laboratory value is before or the same as the time of first study drug administration. If any of these times are missing and the date of laboratory value is equal to the date of first study drug administration, then the laboratory assessment will be considered as according to protocol, i.e. as prior to first study medication.

## 7. PLANNED ANALYSIS

For End-Of-Text (EoT) tables, the set of summary statistics is: N / Mean / SD / Min / Q1 (lower quartile) / Median / Q3 (upper quartile) / Max.

Tabulations of frequencies for categorical data will include all possible categories and will display the number of observations in a category as well as the percentage (%) relative to the respective treatment group (unless otherwise specified, all patients in the respective patient set whether they have non-missing values or not). Percentages will be rounded to one decimal place. The category missing will be displayed only if there are actually missing values.

#### 7.1 DEMOGRAPHIC AND OTHER BASELINE CHARACTERISTICS

Only descriptive statistics are planned for this section of the report.

#### 7.2 CONCOMITANT DISEASES AND MEDICATION

Only descriptive statistics are planned for this section of the report.

#### 7.3 TREATMENT COMPLIANCE

Only descriptive statistics are planned for this section of the report.

# 7.4 PRIMARY ENDPOINT(S)

## 7.4.1 Dose Finding Part:

One of the primary objectives is to assess the MTD based on the number of patients presenting DLTs during the MTD evaluation period. Therefore, an overall summary of DLTs (see CTP Section 4, Table 4.1.4.1.2 for the definition of DLTs) which occurred during the MTD evaluation period will be provided for each dose cohort from the dose finding cohort treated set. Patients who were replaced within the MTD evaluation period will be excluded from the determination of the MTD but will be considered for all other safety evaluations.

A summary of the number of patients with DLTs overall in any course will be also given by initial treatment and displayed in a similar format to the summary of DLTs occurring in the MTD evaluation period.

The determination of the MTD is based on a Rolling 6 design as illustrated in Section 4, Table 4.1.4.1:1 of the CTP. The MTD is defined as the highest dose at which no more than 1/6 patients experienced DLT considered related to a fatinib during the MTD evaluation period. Refer to CTP 7.3.1 for further details on MTD evaluation.

Analysis of the standard PK endpoints is performed according to (2) and (8) as outlined in Section 7.3.5 of the CTP.

### 7.4.2 MTD expansion cohort part:

Objective response (OR) is defined as a best overall response of complete response (CR) or partial response (PR) based on investigator's assessment according to the institutional

TSAP for BI Trial No: 1200.120 Proprietary confidential information © 2020 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

response evaluation criteria for the given tumour type. If the International Criteria for Neuroblastoma Response Criteria (INRC) is used, OR is defined as complete response (CR), very good partial response (VGPR), partial response (PR) and mixed response (MxR). For further details on OR, please refer to CTP Section 7.3.1. The objective response rate will be calculated and reported as proportion of responders with 95% Clopper-Pearson CIs based on all treated patients. Objective response will be summarized regardless of confirmation.

Additional summary or listing may be provided for confirmed response. If only few patients (fewer than 5) achieved objective response, a detailed listing will be reported.

For objective responses, evaluated by institutional response evaluation criteria other than INRC, below confirmation rule for best overall response will be considered.

If CR or PR: look at all subsequent visits, if there is another CR or PR >=28 days then the patient has a confirmed response. If there is not another CR or PR >=28 days then the patient can be SD. Please note that once patient achieve CR any response other than CR will be considered as PD.

Detailed specifications are listed in Table 7.4.2: 1.

Table 7.4.2: 1 Confirmation rule for best overall response

| Overall response | Overall response | Unconfirmed best | Confirmed best overall |
|---|---|---|---|
| (time point 1) | (subsequent time point) | overall response | response |
| CR | CR (>=28 days from 1) | CR | CR |
| CR | CR (< 28 days from 1) | CR | SD |
| CR | PR <sup>1</sup> | CR | SD |
| CR | SD | CR | SD |
| CR | PD | CR | SD |
| CR | NE/Missing | CR | SD |
| PR | CR (>=28 days from 1) | CR | PR |
| PR | CR (< 28 days from 1) | CR | SD |
| PR | PR (>=28 days from 1) | PR | PR |
| PR | PR (< 28 days from 1) | PR | SD |
| PR | SD | PR | SD |
| PR | PD | PR | SD |
| PR | NE/Missing | PR | SD |

<sup>1=</sup> If truly a CR at first response, any subsequent disease (even a PR relative to baseline) makes the disease PD. Could only be a PR if initial CR is changed to PR (i.e. not a true CR).

For INRC, a similar derivation of confirmed response will apply. That is, a subsequent assessment with the same or a better overall response on or after 28 days is required for the confirmation of an objective response, in the order from best to worst of CR > VGPR > PR > MxR. Otherwise, a SD will be considered as the confirmed best overall response.

#### 7.5 SECONDARY ENDPOINT(S)

#### 7.5.1 **Key secondary endpoint(s)**

This section is not applicable as no key secondary endpoint has been specified in the protocol.

# 7.5.2 (Other) Secondary endpoint(s)

For progression free survival (PFS), objective response (OR) and duration of objective response (DoR), a descriptive and graphical summary of the endpoint will be provided. The Kaplan-Meier estimates of PFS and DoR (if applicable) and 95% confidence intervals will be calculated at the time of each planned assessment. For the dose finding part, the number of patients with OR will be summarized by dose level. If fewer than 5 patients achieved OR, then DoR will only be listed; Kaplan-Meier estimates will not be calculated and no summary table or graph will be provided.

To evaluate the potential influence of age on pharmacokinetic parameters like C<sub>max</sub> and AUC, an exploratory subgroup analysis will be performed for different age groups. For this, binning of age into groups will be performed to ensure that groups have reasonable patient numbers. If feasible, a correlation of age and PK parameters may be performed.

### 7.7 EXTENT OF EXPOSURE

Treatment exposure will be primarily summarized by the total on-treatment time and has been defined in <u>Section 5.4</u> of this TSAP.

Treatment interruptions before permanent discontinuation will not be excluded. Summary statistics for treatment time by each dose level of afatinib over time will also be provided.

#### 7.8 SAFETY ANALYSIS

All safety analyses will be performed on the treated set.

### 7.8.1 Adverse events

The analyses of adverse events (AE) will be descriptive in nature. All analyses of AEs will be based on the number of patients with AEs and not on the number of AEs. For analysis of duration, severity etc. of multiple AE occurrences, data on the case report form (CRF) will be collapsed into AE episodes provided that all of the following applies:

- The same MedDRA lowest level term was reported for the occurrences.
- The occurrences were time-overlapping or time-adjacent (time-adjacency of two occurrences is given if the second occurrence started on the same day or on the day after the end of the first occurrence).
- Treatment did not change between the onset of the occurrences or treatment changed between the onsets of the occurrences, but no deterioration was observed for the later occurrence.

For further details on summarization of AE data, please refer to the BI guideline (4).

The analyses of adverse events will be based on the concept of treatment-emergent adverse events. That means that all adverse events occurring between first drug intake and 28 days after last drug intake or death, whichever occurs first, will be assigned to the on-treatment period. All adverse events occurring before any study drug intake will be assigned to 'screening' and all adverse events occurring after last study drug intake + 28 days will be assigned to 'Off-treatment' (for listings only). For details on the treatment definition, see Section 6.1.

An overall summary of adverse events will be presented. The frequency of patients with adverse events will be summarised by highest CTC grade (grades 1, 2, 3, 4, 5 and all grades), treatment, primary system organ class and preferred term for each of the following AE tables as well as relatedness of AEs to treatment and seriousness:

- DLTs (1<sup>st</sup> course and all courses)
- All AEs
- Drug-related AEs
- AEs leading to dose reduction
- AEs leading to treatment discontinuation
- Drug-related AEs leading to dose reduction
- Drug-related AEs leading to treatment discontinuation
- AEs leading to death
- Serious AEs
- Drug related serious AEs
- Other significant AEs, defined as AEs leading to dose reduction or permanent discontinuation of study medication
- Non-serious AEs with higher than 5% occurrence rate for disclosure on ClinicalTrials.gov

Please refer to CTP Section 5.2.2.1 for definitions of the adverse events. All tables will be sorted by system organ classes (SOC) according to the standard sort order specified by the European Medicines Agency (EMA). Preferred terms (PTs) will be sorted by frequency (within SOC).

The table for all AEs will be repeated with the project defined grouping of AE terms (acute renal failure associated with severe diarrhoea, acne, rash, stomatitis, conjunctivitis, paronychia, severe cutaneous adverse reactions, interstitial lung disease, keratitis, hepatic impairment, pancreatitis, heart failure, gastrointestinal perforation, hypersensitivity reactions, nail disorders and fatigue). Details of the project defined groupings will be defined in the technical TSAP. In these tables the grouped AEs will replace the original PTs for all AEs that are included within the grouped term. The grouped AE categories will then be tabulated along with all remaining MedDRA PTs, sorted by descending frequency.

A reference table presenting the entire project defined groupings and MedDRA PTs within each grouping will also be produced.

Additional AE tables will be produced for AEs of special interest (hepatic injury as defined in CTP Section 5.2.2.1 and dose limiting toxicities as defined by CTP Section 4, table 4.1.4.2). Listings providing further details on highest CTC grade, action taken with study drug and time to first onset of AE will be produced.

### 7.8.2 Laboratory data

The analyses of laboratory data will be descriptive in nature and will be based on BI standards (5). The same on-treatment period as considered for the analysis of AEs will be applied for laboratory values. CTC grade for applicable lab parameters will be calculated according to CTCAE v3.0 (7).

For a list of laboratory parameters considered for this trial, please refer to CTP Section 5.2.3, Table 5.2.3:1. Descriptive statistics of all normalized laboratory values by visit will be provided including changes from baseline. Transition tables of CTCAE grade from baseline to worst value and last value on treatment, and frequency tables of possible clinically significant abnormalities will be produced. For those parameters that have CTC grading possible clinically significant abnormalities are defined as those laboratory values with a CTC grade  $\geq$  2 that have had an increase of  $\geq$  1 grade from baseline. For those parameters for which no CTC grade has been defined standard BI project definitions will be used to decide on clinical significance. See Tables 7.8.2: 1 and 7.8.2: 2 for the potential clinical significance rules.

Analyses of descriptive statistics will use normalized lab values (variables ULN, LABN). Analyses of frequencies of patients with potential clinical significance, analyses of shift, and liver function categories tables will use converted values (ULC, LABSTD).

Summaries will be produced of laboratory data recorded on-treatment. Listings will be provided for data recorded prior to treatment, on-treatment and post-treatment. For details on the treatment definition, see Section 6.1.

For the primary laboratory parameters listed in Table 7.8.2: 1, full analysis of descriptive statistics, transition tables and possible clinical significant abnormalities will be conducted.

Analysis of secondary laboratory parameters listed in <u>Table 7.8.2: 2</u> will be limited to frequency tables of possible clinically significant abnormalities. Listings of converted and normalized values for all laboratory parameters considered for this trial will be provided in Appendix 16.2 of the CTR.

Table 7.8.2: 1 Primary laboratory parameters

| Label | Lab test name | Direction of interest | Potential clinical significance rule |
|---|---|---|---|
| ALKP | Alkaline phosphatase | High | $A^1$ |
| APTT | APTT (Activated partial thrombopl. time) | High | $A^1$ |
| CRE | Creatinine | High | A <sup>1</sup> |
| CRECL | GFR/Creatinine clearance | Low | $A^{1,2}$ |
| HGB | Haemoglobin | Low | A <sup>1</sup> |
| INR | PT-INR | High | $A^1$ |
| K | Potassium | Low | $A^1$ |
| LYMPH | Lymphocytes | Low | A <sup>1</sup> |
| NA | Sodium | Low | A <sup>1</sup> |
| NEUT | Neutrophils | Low | $A^1$ |
| SGOT | AST/GOT, SGOT | High | A <sup>1</sup> |
| SGPT | ALT/GPT, SGPT | High | $A^1$ |
| TBILI | Bilirubin, total | High | $A^1$ |
| WBC | White blood cell ct. | Low | $A^1$ |

<sup>&</sup>lt;sup>1</sup>A = CTCAE grade 2 or greater with an increase of at least one CTCAE grade from baseline. <sup>2</sup>Values less than 0.25xLLN will be assigned CTCAE grade 3.

Table 7.8.2: 2 Secondary laboratory parameters

| Label | Lab test name | Direction of interest | Potential clinical significance rule |
|---|---|---|---|
| BUN | Blood urea nitrogen | High | > 10 |
| CA | Calcium | Low & High | $A^1$ |
| CK | Creatine kinase | High | $A^1$ |
| GLUB | Glucose | Low & High | $A^1$ |
| LDH | LDH | High | ≥3xULN |
| TPRO | Protein, total | Low & High | < 45, > 100 |
| UREA | Urea | High | > 1.5xULN |
| URIC | Uric acid | High | $A^{1,3}$ |

A = CTCAE grade 2 or greater with an increase of at least one CTCAE grade from baseline.  $^{3}$ Values >ULN – 10 mg/dL or  $\leq$ 0.59 mmol/L will be assigned CTCAE grade 1.

#### 7.8.3 Vital signs

Only descriptive statistics are planned for this section of the report.

#### 7.8.4 **ECG**

ECG data will be collected as described in CTP Section 5.2.4. Clinically significant findings in ECG data will be reported under "Adverse events" if applicable and will be analysed accordingly.

#### 7.8.5 **Others**

# Left ventricular ejection function:

Left ventricular ejection function (LVEF) will be assessed by echocardiography (ECHO) as specified in the CTP Section 5.2.5.2.

### Attainment of steady-state:

Attainment of steady-state will be assessed graphically.

TSAP for BI Trial No: 1200.120 Proprietary confidential information © 2020 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 8. **REFERENCES**

| 1 | CPMP/ICH/363/96: "Statistical Principles for Clinical Trials", ICH Guideline Topic E9, |
|---|---|
| | Note For Guidance on Statistical Principles for Clinical Trials, current version. |
| 2 | 001-MCS 36-472: "Standards and processes for analyses performed within Clinical |
| | Pharmacokinetics/Pharmacodynamics", current version; KMED |
| 3 | BI-KMED-BDS-HTG-0035: "Handling of Missing and Incomplete AE Dates", current |
| | version; KMED |
| 4 | BI-KMED-BDS-HTG-0066: "Analysis and Presentation of Adverse Event Data from |
| | Clinical Trials", current version; KMED |
| 5 | BI-KMED-BDS-HTG-0042: "Handling, Display and Analysis of Laboratory Data", |
| | current version; KMED |
| 6 | BI-KMED-BDS-QRG-0011: "BI Lab Standards", current version; KMED |
| 7 | Common Terminology Criteria for Adverse Events (CTCAE) Version 3.0, published: |
| | August 9, 2006; U.S. Department of Health and Human Services, National Institutes of |
| | Health, National Cancer Institute. |
| 8 | BI Position Paper 3.8: Statistical Methods for PK, current version. |

# **Boehringer Ingelheim**

TSAP for BI Trial No: 1200.120 Proprietary confidential information © 2020 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

TSAP for BI Trial No: 1200.120 

Proprietary confidential information © 2020 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### **10. HISTORY TABLE**

This is a revised TSAP including the following modifications to the final TSAP.

Table 10: 1 History table

| Version | Date | Author | Sections | Brief description of change |
|---|---|---|---|---|
| | (DD-MMM-YY) | | changed | |
| Final | 17-JAN-18 | | None | This is the final TSAP without any |
| | | | | modification |
| Revised | 14-JUL-20 | | All | |
| | | | | dded |
| | | | | disease control as additional secondary endpoint. |
| | | | | enapoint. |
| | | | | Section 5: Aligned endpoint definitions |
| | | | | with protocol. Added censoring rules for |
| | | | | PFS. |
| | | | | Section 6: Clarified definitions of |
| | | | | analysis treatment periods. Updated |
| | | | | definitions of important protocol |
| | | | | deviation. Updated definition of PK |
| | | | | analysis set. |
| | | | | Section 7: Added confirmation rule for |
| | | | | best overall response. Clarified analysis |
| | | | | of DoR when number of patients with OR is low. |
| | | | | Updated analysis plan |
| | | | | for adverse events and safety laboratory |
| | | | | data. Added attainment of steady state |
| | | | | analysis. |
| | | | | Section 8: Updated references to current |
| | | | | company guidelines. |
| Revised | 31-JUL-20 | | Sections | The definition of "Duration of objective |
| 1001000 | 01-00L-20 | | 4 and | response", a secondary endpoint, was |
| | | | 5.2.2 | incorrect in the CTP. A clarification is |
| | | | | added in Section 4. The correct |
| | | | | definition is provided in Section 5.2.2. |